CLINICAL TRIAL: NCT02909452
Title: A Phase 1, Randomized, Open-Label, Continuation Study of Entinostat in Combination With Pembrolizumab in Patients With Advanced Solid Tumors (SNDX-275-0141, MK3475-460/KEYNOTE-460)
Brief Title: Continuation Study of Entinostat in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0141
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Breast Diseases; Renal Neoplasm; Solid Tumors
Keywords: entinostat; pembrolizumab; solid tumor; Histone Deacetylase Inhibitor
MeSH Terms: conditions — Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Breast Diseases; Kidney Neoplasms | interventions — entinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ENT 1mg daily with pembro every 3 weeks (Active Comparator): Entinostat daily in combination with pembrolizumab every three weeks
  Interventions: Drug: Entinostat; Drug: Pembrolizumab
- ENT 5mg weekly with pembro every 3 weeks (Active Comparator): Entinostat once weekly in combination with pembrolizumab every three weeks
  Interventions: Drug: Entinostat; Drug: Pembrolizumab
- ENT 10mg bi-weekly with pembro every 3 weeks (Active Comparator): Entinostat once every other week in combination with pembrolizumab every three weeks
  Interventions: Drug: Entinostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Entinostat — HDAC (histone deacetylase) inhibitor
  Other Names: SNDX-275; MS-275
Drug: Pembrolizumab — A selective humanized monoclonal antibody (mAb)
  Other Names: Keytruda; MK-3475; SCH-900475

SUMMARY:
The objectives of this study are to explore different dosing levels and schedules of entinostat in combination with pembrolizumab in patients with advanced solid tumors, in terms of safety, tolerability, pharmacokinetics (PK), impact on immune correlatives, and efficacy

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single center, randomized study to assess the safety and tolerability of 3 different dose regimens of entinostat in combination with pembrolizumab in patients with advanced solid tumors who previously completed Study SNDX-275-0140 (NCT02897778). Up to 30 patients will be randomized in a 1:1:1 fashion to one of three arms. In the event that greater than or equal to 2 out of the first 6 patients randomized experience a dose-limiting toxicity, the next patient randomized to that Arm will receive treatment at a reduced starting dose as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Completed Study SNDX-275-0140 (NCT02897778)
2. Any AE or toxicity experienced in Study SNDX-275-0140 (NCT02897778) is resolved to less than or equal to Grade 1
3. Continues to meet inclusion criteria for Study SNDX-275-0140 (NCT02897778) at the time of entry into this study

Exclusion Criteria:

1. Completed Study SNDX-275-0140 (NCT02897778) more than 30 days prior to Cycle 1 Day 1 of this study
2. Continues to meet exclusion criteria for Study SNDX-275-0140 (NCT02897778) at the time of entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events (AEs) resulting in the permanent discontinuation of study drug, and deaths occurring within the reporting period required for the study | Each treatment cycle is 21 days. All events will be collected from informed consent through 90 days post-last dose or through 30 days after initiation of new anti-cancer therapy
Changes from baseline in laboratory results | Baseline through 90 day safety follow-up visit
Changes from baseline in vital signs | Baseline through 90 day safety follow-up visit
Changes from baseline in ECG results | Baseline through 90 day safety follow-up visit

SECONDARY OUTCOMES:
AUC0-t (area under the curve to last observed concentration time) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1
AUC0-inf (area under the curve extrapolated to infinity) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1
Cmax (maximum plasma concentration) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1
Tmax (time to maximum plasma concentration) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1
T1/2 (elimination half life) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1
Vd (clearance and volume of distribution) of entinostat when given in combination with pembrolizumab | Pre-dose through Cycle 3 Day 1

OTHER OUTCOMES:
Ratio of effector T cells to regulatory T cells in blood pre-therapy and post-therapy | Pre-dose through Cycle 3 Day 1
Changes in the number of circulating immune related cells | Pre-dose through Cycle 3 Day 1
Changes in protein lysine acetylation in peripheral blood cells pre-therapy and post-therapy | Pre-dose through Cycle 3 Day 1
Best overall tumor response | Baseline up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meyers, MD, PhD, Study Director — Syndax Pharmaceuticals
Locations (1):
- The START Center for Cancer Care, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reviewed throughout the study by the sponsor, clinical research organization assisting with SAE management, and routine monitoring to safeguard the interests of the trial patients and to assess the safety of the interventions administered during the trial.